CLINICAL TRIAL: NCT04443972
Title: Evaluation of Injectable Beta- Tricalcium Phosphate as an Occlusive Barrier Membrane in Treatment of Grade ii Furcation Involvement (Clinical and Radiographic Study)
Brief Title: Evaluation of Injectable Beta-tricalcium Phosphate Clinically in Treatment of Grade II Furcation Involvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Furcation invlvement
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Furcation Defects
Keywords: Grade II Furcation defects
MeSH Terms: conditions — Furcation Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD VitalOs cement® alone (Experimental): class II furcation defects that will be treated with PD VitalOs cement® alone
  Interventions: Other: PD VitalOs cement®
- PD VitalOs cement® plus Bone graft and membrane (Experimental): PD VitalOs cement® and Hydroxyapatite bone graft and biodegradable collagen membrane in the treatment of class II furcation defects.
  Interventions: Other: PD VitalOs cement®; Other: Hydroxyapatite bone graft; Other: biodegardable collagen membrane

INTERVENTIONS:
Other: PD VitalOs cement® — PD VitalOs cement®* is a synthetic bone grafting cement designed for bone void filling and bone regeneration in dental surgery
Other: Hydroxyapatite bone graft — a bioceramic bone substitute, providing a scaffold for bone deposition
  Arms: PD VitalOs cement® plus Bone graft and membrane
Other: biodegardable collagen membrane — provide efficacious barriers that were interposed between the flap and root surface.
  Arms: PD VitalOs cement® plus Bone graft and membrane

SUMMARY:
This study will be conducted to evaluate clinically and radiographically the use of PD VitalOs cement® bone graft in the treatment of class II furcation defects comparing with Hydroxyapatite bone graft and biodegradable collagen membrane in the treatment of class II furcation defects.

DETAILED DESCRIPTION:
The study is a randomized, controlled clinical trial. Patients were randomly divided into two equal groups, Group I (Test group): included seven Grade II furcation defects treated by beta tricalcium phosphate bone cement only.

Group II (Control group): included seven Grade II furcation defects treated with granulated beta tricalcium phosphate bone graft covered by resorbable collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* • Presence of a lower molar with critical size grade II furcation defect (15) with a horizontal component of 4 mm and a vertical component of 4 to 6 mm (18), detected using Naber's probe and William's periodontal probe.

  * Patient's age between 30 - 50 years.
  * Both sexes.
  * The patient should be psychologically accepting the procedures.
  * Patients should be systemically free.

Exclusion Criteria:

* • Uncooperative patients regarding oral hygiene measures performance.

  * Patients with para functional habits.
  * Smokers.
  * Pregnant or lactating women.
  * Patients who underwent any periodontal surgeries in the study site during the six months prior to study.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
change in plaque index scores (PI) according to Silness and Löe. | at 3 weeks and 6 weeks
  Score 0 = no plaque in gingival area. Score 1= film of plaque adhering to the free gingival margin and the adjacent area of the tooth, plaque may only be recognized by running a probe across the tooth surface.
  Score 2= moderate accumulation of soft deposits within the gingival pocket and on the gingival margin and/ or adjacent tooth surface which can be seen by the naked eye.
  Score 3= abundant of soft matter within gingival pocket and/ or the gingival margin and adjacent tooth surface.
  The scores from the four surfaces of the tooth were added and divided by (four) to give plaque index for each tooth; the plaque index score for an individual was obtained by adding the indices of the teeth and dividing by the number of the teeth examined.
change in probing Pocket Depth(PPD) | at 3 weeks and 6 weeks
  The measurements were carried out to the defects selected using an 0.8 mm thick periodontal probe * with William's calibration, which was marked from (1-10) mm, pocket depth of (1 mm) or less was recorded as (1mm),measurements exceeding (1mm) but less than (2mm) were recorded as (2mm) so that the probing pocket depth was measured to the nearest mm.
  Probing pocket depth refers to the distance from the gingival margin to the bottom of the pocket. Mesial and distal pockets were measured as well as the furcation from the buccal aspect as close as possible to the contact points, facial and lingual pockets were measured at midline of roots.
  Efforts were made to insert the probe parallel to the long axis of the roots. Light force was used during the introduction of the probe to the bottom of the pocket, third molars and teeth with enamel projections were excluded. (7)
change in clinical Attachment Level | at 3 weeks and 6 weeks
  The measurements were carried out to the defects selected using an 0.8 mm thick periodontal probe * with William's calibration, which was marked from (1-10) mm, pocket depth of (1 mm) or less was recorded as (1mm),measurements exceeding (1mm) but less than (2mm) were recorded as (2mm) so that the probing pocket depth was measured to the nearest mm.
  Probing pocket depth refers to the distance from the gingival margin to the bottom of the pocket. Mesial and distal pockets were measured as well as the furcation from the buccal aspect as close as possible to the contact points, facial and lingual pockets were measured at midline of roots.
  Efforts were made to insert the probe parallel to the long axis of the roots. Light force was used during the introduction of the probe to the bottom of the pocket, third molars and teeth with enamel projections were excluded. (7)

SECONDARY OUTCOMES:
change in radiographic bone level (RBL) | at basline, 3 and 6 months
change in optical density(OD) | at basline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hosny Elsayed, BDS, Principal Investigator — Alexandria University; shahira Ali El Damaty, PHD, Study Director — Alexandria University; Gehan Sherif Kotry, PHD, Study Director — Alexandria University; Rania Abd El Aziz Fahmy, PHD, Study Director — Alexandria University
Locations (1):
- outpatient clinic of oral medicine department, faculty of dentistry, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutando A, Galindo P, Gomez-Moreno G, Arana C, Bolanos J, Acuna-Castroviejo D, Wang HL. Relationship between salivary melatonin and severity of periodontal disease. J Periodontol. 2006 Sep;77(9):1533-8. doi: 10.1902/jop.2006.050287. PMID 16945031
- [Background] Bowers GM, Schallhorn RG, McClain PK, Morrison GM, Morgan R, Reynolds MA. Factors influencing the outcome of regenerative therapy in mandibular Class II furcations: Part I. J Periodontol. 2003 Sep;74(9):1255-68. doi: 10.1902/jop.2003.74.9.1255. PMID 14584858
- [Background] Laurell L, Gottlow J, Zybutz M, Persson R. Treatment of intrabony defects by different surgical procedures. A literature review. J Periodontol. 1998 Mar;69(3):303-13. doi: 10.1902/jop.1998.69.3.303. PMID 9579616
- [Background] Nasr HF, Aichelmann-Reidy ME, Yukna RA. Bone and bone substitutes. Periodontol 2000. 1999 Feb;19:74-86. doi: 10.1111/j.1600-0757.1999.tb00148.x. PMID 10321217
- [Background] Caton JG. Overview of clinical trials on periodontal regeneration. Ann Periodontol. 1997 Mar;2(1):215-22. doi: 10.1902/annals.1997.2.1.215. PMID 9151555
- [Background] Mendieta C, Williams RC. Periodontal regeneration with bioresorbable membranes. Curr Opin Periodontol. 1994:157-67. PMID 8032456
- [Background] Gray JL, Hancock EB. Guided tissue regeneration. Nonabsorbable barriers. Dent Clin North Am. 1998 Jul;42(3):523-41. PMID 9700453
- [Background] Baum BJ, Mooney DJ. The impact of tissue engineering on dentistry. J Am Dent Assoc. 2000 Mar;131(3):309-18. doi: 10.14219/jada.archive.2000.0174. PMID 10715922
- [Background] Cury PR, Sallum EA, Nociti FH Jr, Sallum AW, Jeffcoatt MK. Long-term results of guided tissue regeneration therapy in the treatment of class II furcation defects: a randomized clinical trial. J Periodontol. 2003 Jan;74(1):3-9. doi: 10.1902/jop.2003.74.1.3. PMID 12593590
- [Background] Basten CH, Ammons WF Jr, Persson R. Long-term evaluation of root-resected molars: a retrospective study. Int J Periodontics Restorative Dent. 1996 Jun;16(3):206-19. PMID 9084307
- [Background] Hamp SE, Nyman S, Lindhe J. Periodontal treatment of multirooted teeth. Results after 5 years. J Clin Periodontol. 1975 Aug;2(3):126-35. doi: 10.1111/j.1600-051x.1975.tb01734.x. PMID 1058213
- [Background] Hirschfeld L, Wasserman B. A long-term survey of tooth loss in 600 treated periodontal patients. J Periodontol. 1978 May;49(5):225-37. doi: 10.1902/jop.1978.49.5.225. PMID 277674
- [Background] Kenney EB, Lekovic V, Elbaz JJ, Kovacvic K, Carranza FA Jr, Takei HH. The use of a porous hydroxylapatite implant in periodontal defects. II. Treatment of Class II furcation lesions in lower molars. J Periodontol. 1988 Feb;59(2):67-72. doi: 10.1902/jop.1988.59.2.67. PMID 2831333
- [Background] Eickholz P, Hausmann E. Evidence for healing of Class II and Class III furcations 24 months after guided tissue regeneration therapy: digital subtraction and clinical measurements. J Periodontol. 1999 Dec;70(12):1490-500. doi: 10.1902/jop.1999.70.12.1490. PMID 10632525
- [Background] De Leonardis D, Garg AK, Pedrazzoli V, Pecora GE. Clinical evaluation of the treatment of class II furcation involvements with bioabsorbable barriers alone or associated with demineralized freeze-dried bone allografts. J Periodontol. 1999 Jan;70(1):8-12. doi: 10.1902/jop.1999.70.1.8. PMID 10052766
- [Background] Ohura K, Bohner M, Hardouin P, Lemaitre J, Pasquier G, Flautre B. Resorption of, and bone formation from, new beta-tricalcium phosphate-monocalcium phosphate cements: an in vivo study. J Biomed Mater Res. 1996 Feb;30(2):193-200. doi: 10.1002/(SICI)1097-4636(199602)30:23.0.CO;2-M. PMID 9019484
- [Background] Flautre B, Lemaitre J, Maynou C, Van Landuyt P, Hardouin P. Influence of polymeric additives on the biological properties of brushite cements: an experimental study in rabbit. J Biomed Mater Res A. 2003 Aug 1;66(2):214-23. doi: 10.1002/jbm.a.10539. PMID 12888990
- [Background] Meikle MC, Papaioannou S, Ratledge TJ, Speight PM, Watt-Smith SR, Hill PA, Reynolds JJ. Effect of poly DL-lactide--co-glycolide implants and xenogeneic bone matrix-derived growth factors on calvarial bone repair in the rabbit. Biomaterials. 1994 Jun;15(7):513-21. doi: 10.1016/0142-9612(94)90017-5. PMID 7918904
- [Background] Miyamoto S, Takaoka K, Okada T, Yoshikawa H, Hashimoto J, Suzuki S, Ono K. Polylactic acid-polyethylene glycol block copolymer. A new biodegradable synthetic carrier for bone morphogenetic protein. Clin Orthop Relat Res. 1993 Sep;(294):333-43. PMID 8358939
- [Background] Aichelmann-Reidy ME, Yukna RA. Bone replacement grafts. The bone substitutes. Dent Clin North Am. 1998 Jul;42(3):491-503. PMID 9700451
- [Background] Melcher AH. On the repair potential of periodontal tissues. J Periodontol. 1976 May;47(5):256-60. doi: 10.1902/jop.1976.47.5.256. No abstract available. PMID 775048
- [Background] Blumenthal NM. A clinical comparison of collagen membranes with e-PTFE membranes in the treatment of human mandibular buccal class II furcation defects. J Periodontol. 1993 Oct;64(10):925-33. doi: 10.1902/jop.1993.64.10.925. PMID 8277399
- [Background] Cortellini P, Prato GP. Guided tissue regeneration with a rubber dam: a five-case report. Int J Periodontics Restorative Dent. 1994 Feb;14(1):8-15. PMID 8005773
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370
- [Background] Garrett S, Martin M, Egelberg J. Treatment of periodontal furcation defects. Coronally positioned flaps versus dura mater membranes in class II defects. J Clin Periodontol. 1990 Mar;17(3):179-85. doi: 10.1111/j.1600-051x.1990.tb01083.x. PMID 2319003
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Glavind L, Loe H. Errors in the clinical assessment of periodontal destruction. J Periodontal Res. 1967;2(3):180-4. doi: 10.1111/j.1600-0765.1967.tb01887.x. No abstract available. PMID 4237475